CLINICAL TRIAL: NCT00931983
Title: The Effect of Locomotor Training on Children With Incomplete Spinal Cord Injuries
Status: Withdrawn | Type: Observational
Sponsor: McGill University (Other)
Collaborators: Rick Hansen Foundation (Other); Shriners Hospitals for Children (Other); Fondation pour la Recherche sur la Moelle Épinière (Spinal Cord Research Foundation) (Unknown)
Responsible Party: Mohan Radhakrishna, Md, FRCSC, Shriners Hospitals for Children-Canada
Other Study IDs: 2009-38
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-07

CONDITIONS: Spinal Cord Injuries
Keywords: Incomplete spinal cord injuries; Walking; Treadmill; Training
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
--Participation open to all Canadian residents--

The purpose of this study is to address how well children with incomplete spinal cord injuries of greater than 12 months duration who remain non-functional ambulators improve through body weight assisted treadmill training (BWATT).

DETAILED DESCRIPTION:
In the past, this type of treatment has been offered to adults living with a spinal cord injury, but only recently has it been extended, in the US, to children so affected. Numerous trials indicate that BWSTT does improve human gait patterns in adults. As children have more neuroplasticity than adults, we believe they should respond well to BWSTT.

The BWSTT uses a counterweight harness system to unload the patient's body weight while he or she is on a treadmill. The patient's legs are manually moved by trained therapists through the human gait cycle while maintaining a correct upright posture. Functional and social re-integration outcome assessments are administered before and after each treatment period.

The aim, this year, is to recruit five children who have been living with a spinal cord injury for at least 12 months. The 12-month timeframe was chosen to limit any gait improvement from spontaneous recovery as well as to ensure medical stability.

The study will be conducted over a nine-week period. There are two three-week training sessions separated by a three-week rest period. The BWSTT therapy will be held twice daily for 30 minute sessions. The children and their families return home between the two training periods and are allowed to continue any conventional physiotherapy program they started prior to participating in the study. Outcomes will be re-evaluated during the second three-week training period.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 4-18 with incomplete ASIA C or D spinal cord injuries at least 12 months before study enrolment
* Non-ambulatory or 'exercise only' ambulators with or without assistive devices
* Normal motor and cognitive development up to time of injury
* Medical Stability

Exclusion Criteria:

* Other neuromuscular disease
* Contraindication to weight bearing on lower extremities
* Pressure sores where harness would be applied
* Uncontrollable hypotension when upright
* Lower limb contractures impeding range of motion necessary for ambulation
* Prior enrolment in a BWATT program
* Unable to commit to intervention for duration of protocol

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-03

PRIMARY OUTCOMES:
10 meter walk | Baseline (time 0)
10 meter walk | 9 weeks

SECONDARY OUTCOMES:
Pediatric Life Habits Questionnaire | baseline (time 0)
Pediatric Life Habits Questionnaire | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Radhakrishna, Md, FRCPC, Principal Investigator — McGill University, Shriners Hospitals for Children-Canada; Hugues Barbeau, Pt, PhD, Study Chair — McGill University; Joanne Ruck-Gibis, Pt, MSc, Study Chair — McGill University; Kathleen Montpetit, Ot, MSc, Study Chair — McGill University, Shriners Hospitals for Children-Canada; Jean Ouellet, Md, FRCSC, Study Chair — McGill University, Shriners Hospitals for Children-Canada
Locations (1):
- Shriners Hospitals for Children-Canada, Montreal, Quebec, Canada

REFERENCES:
- [Background] Barbeau H, Nadeau S, Garneau C. Physical determinants, emerging concepts, and training approaches in gait of individuals with spinal cord injury. J Neurotrauma. 2006 Mar-Apr;23(3-4):571-85. doi: 10.1089/neu.2006.23.571. PMID 16629638
- [Background] Behrman AL, Nair PM, Bowden MG, Dauser RC, Herget BR, Martin JB, Phadke CP, Reier PJ, Senesac CR, Thompson FJ, Howland DR. Locomotor training restores walking in a nonambulatory child with chronic, severe, incomplete cervical spinal cord injury. Phys Ther. 2008 May;88(5):580-90. doi: 10.2522/ptj.20070315. Epub 2008 Mar 6. PMID 18326054